CLINICAL TRIAL: NCT02604680
Title: A Randomized, Controlled Evaluation of the Safety and Efficacy of Topical Treatments for Moderate-Severe Facial Acne Vulgaris
Brief Title: A Safety and Efficacy Evaluation of Topical Treatments for Moderate-Severe Facial Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI1100-203
Record Dates: First submitted 2015-11-12; First posted 2015-11-13 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BLI1100-1 (Experimental): Topical gel
  Interventions: Drug: BLI1100-1
- BLI1100-2 (Experimental): Topical gel
  Interventions: Drug: BLI1100-2
- BLI1100-3 (Experimental): Topical gel
  Interventions: Drug: BLI1100-3
- BLI1100-4 (Experimental): Topical gel
  Interventions: Drug: BLI1100-4
- Placebo (Placebo Comparator): Topical gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLI1100-1 — BLI1100-1 Topical gel
  Arms: BLI1100-1
Drug: BLI1100-2 — BLI1100-2 Topical gel
  Arms: BLI1100-2
Drug: BLI1100-3 — BLI1100-3 Topical gel
  Arms: BLI1100-3
Drug: BLI1100-4 — BLI1100-4 Topical gel
  Arms: BLI1100-4
Drug: Placebo — Placebo - Topical gel
  Arms: Placebo

SUMMARY:
The objective of the study is to compare the safety and efficacy of multiple formulations of BLI1100 to a control group and placebo in treating patients with moderate-severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 12 to 45 years of age, inclusive, in good general health.
2. Clinical diagnosis of facial acne vulgaris
3. Patients with an Investigator's Global Assessment severity score of at least 3 that meet the following lesion count criteria:

   * A minimum of 20 but not more than 50 inflammatory lesions (including the nose)
   * A minimum of 30 but not more than 100 non-inflammatory lesions on the face (including the nose)
   * No nodules are allowed on the entire face.
4. Each patient or parent/guardian will read and sign the consent form as required by IRB regulations. Patients under the age of 18, but of sufficient age to provide assent (as determined by IRB regulations), will complete an assent form.
5. Female patients of childbearing potential must have a negative urine pregnancy test prior to receiving study medication.
6. Treatment with estrogens, androgens, or anti-androgenic agents for a non-contraceptive indication must be stable for 6 months prior to the first dose of study product and remain unchanged during the study.
7. Patients who are willing and able to follow all study procedures, attend all scheduled visits, and successfully complete the study.
8. Patients who are mentally competent in the Investigator's judgment, to provide informed consent/assent to participate in the study

Exclusion Criteria:

1. Patients who had been treated with:

   * systemic retinoids during a 6-month period before Visit 1 or by systemic antibiotics during a 4-week period before Visit 1
   * or by a topical treatment (eg, antibiotics, benzoyl peroxide, retinoids, azelaic acid, resorcinol, salicylates, sulfacetamide sodium and derivatives, glycolic acid, dapsone) or systemic corticosteroids during a 2-week period before the first dose of study medication.
2. History of hereditary angio-edema
3. Pregnancy, lactation or patient, who is not practicing effective contraception.
4. Any clinically relevant finding at their baseline physical examination or dermatological medical history such as severe systemic diseases or diseases of the facial skin.
5. A known endocrine malfunction (hyperthyroidism, hypothyroidism, diabetes, adrenal insufficiency).
6. Erythroderma, immunodeficiency disorders and Mycosis Fungoides
7. History of Epilepsy or Parkinson's disease
8. History of alcohol and/or drug abuse within 5 years of screening
9. Facial hair (beard), excessive scarring, sunburn or other disfigurement that may obscure the accurate assessment of acne grade
10. Any single facial skin condition assessment graded as "Severe" at Visit 1
11. Using drugs known to be photosensitizers because of the possibility of increased phototoxicity.
12. Refusal to cease using the following types of facial products: astringents, toners, abradants, facials, loofahs, peels containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide (BPO), hydroquinone, sulfacetamide sodium or salicylic acid, non-mild facial cleansers, or moisturizers that contain retinol, salicylic acid, or α- or β-hydroxy acids .
13. Using medications that are reported to exacerbate acne .
14. Have had a facial procedure (chemical or laser peel, microdermabrasion, artificial ultraviolet therapy) performed by an esthetician, beautician, physician, nurse, or other practitioner, during the 4 weeks prior to Visit 1.
15. Unwilling to avoid excessive swimming and sun exposure to include artificial UV light exposure (tanning beds).
16. Patients using comedogenic makeup.
17. Have a known hypersensitivity or previous allergic reaction to any of the components .
18. Employees of the clinical research site or organization involved in the study, or an immediate family member (partner, offspring, parents, siblings, or sibling's offspring) of an employee.
19. Have a member of the same household in this trial.
20. Patients who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
21. Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures
22. Patients who withdraw consent before completion of Visit 1 procedures

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 509 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in total lesion count | 12 weeks
Treatment success based on Investigator Global Assessment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (50):
- United States (50):
  - BLI Research Site 27, Birmingham, Alabama
  - BLI Research Site 24, Mobile, Alabama
  - BLI Research Site 51, Tucson, Arizona
  - BLI Research Site 40, Rogers, Arkansas
  - BLI Research Site 57, Chula Vista, California
  - BLI Research Site 56, Costa Mesa, California
  - BLI Research Site 18, Encino, California
  - BLI Research Site 7, Fremont, California
  - BLI Research Site 45, Upland, California
  - BLI Research Site 41, Denver, Colorado
  - BLI Research Site 39, Wheat Ridge, Colorado
  - BLI Research Site 19, Hialeah, Florida
  - BLI Research Site 49, Jupiter, Florida
  - BLI Research Site 12, Miami, Florida
  - BLI Research Site 54, Miami Lakes, Florida
  - BLI Research Site 20, Ormond Beach, Florida
  - BLI Research Site 59, Port Saint Lucie, Florida
  - BLI Research Site 15, St. Petersburg, Florida
  - BLI Research Site 1, Tampa, Florida
  - BLI Research Site 29, Tampa, Florida
  - BLI Research Site 28, Wellington, Florida
  - BLI Research Site 43, West Palm Beach, Florida
  - BLI Research Site 11, Plainfield, Indiana
  - BLI Research Site 33, Louisville, Kentucky
  - BLI Research Site 34, Beverly, Massachusetts
  - BLI Research Site 42, Quincy, Massachusetts
  - BLI Research Site 37, Fort Gratiot, Michigan
  - BLI Research Site 9, Omaha, Nebraska
  - BLI Research Site 47, Omaha, Nebraska
  - BLI Research Site 5, Newington, New Hampshire
  - BLI Research Site 46, Stony Brook, New York
  - BLI Research Site 50, High Point, North Carolina
  - BLI Research Site 52, Wilmington, North Carolina
  - BLI Research Site 32, Cincinnati, Ohio
  - BLI Research Site 55, Norman, Oklahoma
  - BLI Research Site 4, Gresham, Oregon
  - BLI Research Site 60, Philadelphia, Pennsylvania
  - BLI Research Site 10, Johnston, Rhode Island
  - BLI Research Site 53, Goodlettsville, Tennessee
  - BLI Research Site 58, Murfreesboro, Tennessee
  - BLI Research Site 14, Nashville, Tennessee
  - BLI Research Site 30, Beaumont, Texas
  - BLI Research Site 6, Bryan, Texas
  - BLI Research Site 3, Houston, Texas
  - BLI Research Site 8, New Braunfels, Texas
  - BLI Research Site 44, Pflugerville, Texas
  - BLI Research Site 16, San Antonio, Texas
  - BLI Research Site 21, Salt Lake City, Utah
  - BLI Research Site 26, Norfolk, Virginia
  - BLI Research Site 25, Spokane, Washington